CLINICAL TRIAL: NCT00622518
Title: Ear Drops for Children With Otitis Media
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Standard Homeopathic Company (Industry)
Responsible Party: James A. Taylor, MD, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 33097-B; 07-9092-B 01
Record Dates: First submitted 2008-02-13; First posted 2008-02-25 (Estimated); Results first posted 2010-12-02 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2010-11

CONDITIONS: Acute Otitis Media
Keywords: otitis media; children
MeSH Terms: conditions — Otitis Media

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): homeopathic ear drops in addition to standard care for otitis media
  Interventions: Drug: Hyland's earache drops
- 2 (No Intervention): No ear drops, standard care for otitis

INTERVENTIONS:
Drug: Hyland's earache drops — 3-4 drops in affected ear 3 times a day as needed for up to 5 days
  Arms: 1

SUMMARY:
The purpose of this study is to determine if a commercially available homeopathic ear drop preparation is effective in reducing symptoms in children 6 months - 11 years old with acute otitis media. A total of 120 study patients with otitis media will be randomized to receive homeopathic ear drops, or no ear drops, in addition to receiving standard care. It is postulated that children using the ear drops will have more rapid resolution of symptoms and need fewer antibiotics than those randomized to not receive the ear drops.

ELIGIBILITY:
Inclusion Criteria:

* Presenting to participating clinic with otitis media
* Diagnosed with acute otitis media
* Parents rate symptoms as a "moderate problem" or more

Exclusion Criteria:

* Diagnosis of otitis media within preceding 30 days
* Receipt of antibiotics within 2 days
* Perforated ear drum or bullous lesion
* Receipt of homeopathic treatment within 30 days

Ages: 6 Months to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 119 (Actual)
Dates: Start 2008-02; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James A Taylor, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center-Roosevelt Pediatric Care Center, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients were recruited from 2/4/08 through 2/23/09 at a pediatric primary care clinic at the time of a visit for acute otitis media
Groups:
- Ear Drops Plus Standard Therapy: homeopathic ear drops in addition to standard care for otitis media
- Standard Therapy Alone: No ear drops, standard care for otitis including antibiotics and/or medications to help with ear pain including acetaminophen and ibuprofen
Period: Overall Study
Arm/Group | Ear Drops Plus Standard Therapy | Standard Therapy Alone
Started | 59 | 60
Completed | 59 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ear Drops Plus Standard Therapy | Standard Therapy Alone | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 59 | 60 | 119
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 3.6 (2.5) | 3.4 (2.4) | 3.5 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 25 | 55
  Male | 29 | 35 | 64
Region of Enrollment [Number; unit: participants]
  United States | 59 | 60 | 119

OUTCOME MEASURES:

1. Primary Outcome: Resolution of Otitis Media Symptoms
Description: Mean scores as measured on the Ear Treatment Group-5 scale. This scale quantifies severity of symptoms in children with otitis media. There are 5 components to the scale: fever, earache or tugging, feeding, irritability and sleep. For each component symptoms are rated as 0, 4 or 7 based on severity, with higher scores indicating more sever symptoms. For the primary outcome, the scores for each component were summed to determine an overall Ear Treatment Group -5 Scale score. Total scores range from 0-35. Two assessessments were conducted each day.
Time Frame: 5 days
Population: Data were analyzed on participants from whom data diaries were returned and who had data for an assessment. Data were analyzed on the following number of children at each assessment: 1- 50 standard care (SC),40 ear drop (ED) 2- 40SC 35ED 3- 49SC 37ED 4- 40SC 36ED 5- 44SC 35ED 6- 42SC 34ED 7- 44SC 34ED 8- 43SC 31ED 9- 44SC 33ED 10- 44SC 29ED
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ear Drops Plus Standard Therapy | Standard Therapy Alone
Number analyzed (Participants) | 44 | 50
units on a scale
  Assessment 1: day 1, am | 14.2 (8.2) | 16.5 (8.2)
  Assessment 2: day 1, pm | 7.5 (10.5) | 14.1 (7.4)
  Assessment 3: day 2, am | 6.1 (6.7) | 10.8 (8.1)
  Assessment 4: day 2, pm | 6.7 (6.0) | 8.7 (7.8)
  Assessment 5: day 3, am | 6.1 (6.6) | 7.0 (8.3)
  Assessment 6: day 3, pm | 5.2 (6.3) | 7.3 (8.7)
  Assessment 7: day 4, am | 3.8 (6.1) | 5.8 (7.8)
  Assessment 8: day 4, pm | 3.3 (5.1) | 3.7 (5.7)
  Assessment 9: day 5, am | 2.8 (5.7) | 3.7 (5.7)
  Assessment 10: day 5, pm | 2.3 (4.1) | 3.4 (5.7)
Statistical Analysis 1: Comparison: Ear Drops Plus Standard Therapy vs Standard Therapy Alone; Test type: Superiority or Other; p = .002, linear mixed model — P value is based on rating*group interaction term

2. Secondary Outcome: Side Effects of Therapy
Time Frame: 5 days
Population: Specific side effects were collected on patients whose parents returned study diaries (44 from ear drop group and 50 from standard care only group). In addition, parents were telephoned and asked about any serious side effects.
Measure: Number; unit: participants
Arm/Group | Ear Drops Plus Standard Therapy | Standard Therapy Alone
Number analyzed (Participants) | 59 | 60
participants
  Any side effect reported in diary | 29 | 37
  vomiting reported at least once in diary | 5 | 10
  rash reported at least once in diary | 3 | 5
  diarrhea reported at least once in diary | 3 | 12
  "hyper" behavior reported at least once in diary | 3 | 11
  headache reported at least once in diary | 7 | 6
  lethargy reported at least once in diary | 13 | 15
  other symptom reported at least once in diary | 19 | 22
  serious side effect reported | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: The main source of adverse event information was from symptom logs. In addition, parents were asked about significant adverse events during phone calls 12-15 days after enrollment.
Arm/Group | Ear Drops Plus Standard Therapy | Standard Therapy Alone
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/60
Other Adverse Events (participants affected / at risk) | 29/44 | 37/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ear Drops Plus Standard Therapy (N=44) | Standard Therapy Alone (N=50)
vomiting (Gastrointestinal disorders) | 5 | 10
rash (Skin and subcutaneous tissue disorders) | 3 | 5
diarrhea (Gastrointestinal disorders) | 3 | 12
"hyper" behavior (General disorders) | 3 | 11
headache (General disorders) | 7 | 6
lethargy (General disorders) | 13 | 25
other (General disorders) | 19 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No